CLINICAL TRIAL: NCT07159854
Title: TeleRehabilitation: an Innovative User-centered STrategic Approach for the treatMent of Central and Peripheral Neurological sEquelae From Chemotherapy - TRUST_ME
Brief Title: Telerehabilitation in Central and Peripheral Neurological Sequelae From Chemotherapy
Acronym: TRUST_ME
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Fondazione Don Carlo Gnocchi Onlus (Other)
Collaborators: Astir S.r.l. (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: TRUST_ME
Record Dates: First submitted 2025-08-29; First posted 2025-09-08 (Actual); Last update posted 2025-09-08 (Actual); Status verified 2025-08

CONDITIONS: Chemotherapy-induced Neurotoxicity
Keywords: Chemotherapy-induced neurotoxicity; rehabilitation; telerehabilitation

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- TRUST_ME (Experimental): A cycle of motor and cognitive activities delivered at home through a telerehabilitation approach using the Maia platform by ABmedica (https://abmedica.it/prodotti-ab-medica/maia). The treatment will last 5 weeks with a frequency of three sessions a week (1 synchronous and 2 asynchronous).
  Interventions: Device: RICORDO-DTx system; Device: HOMING system
- Treatment as Usual (Placebo Comparator): Home-based training instructions "as usual", consisting of multimedia content (i.e., videos of the educational/rehabilitation activities) delivered asynchronously via telemedicine platfom. The treatment will last 5 weeks with a frequency of three sessions a week.
  Interventions: Device: Home-based training program

INTERVENTIONS:
Device: RICORDO-DTx system — Participants with will undergo a cognitive enhancement program using the Astir RICORDO-DTx system (http://www.ricordo-dtx.com), which allows for the personalization of rehabilitative content based on the needs of the target population and can be delivered remotely.
  Arms: TRUST_ME
Device: HOMING system — Participants will also undergo motor rehabilitation sessions focused on improving balance, gait, and muscular endurance using the HOMING system (https://www.tecnobody.com/homing).
  Arms: TRUST_ME
Device: Home-based training program — Subjects will view videos on Tablet. The treatment will be provided via a digital medicine platform on a mobile device (tablet).
  Arms: Treatment as Usual

SUMMARY:
The goal of this clinical trial is to validate the use of innovative tele-rehabilitation (TR) models in terms of efficiency and effectiveness in a pilot cohort of subjects with central and peripheral chemotherapy-induced neurotoxicity. Participants will be randomized (with an allocation ratio of 1:1) into the experimental group (TRUST_ME - 15 sessions of motor and cognitive activities delivered at home through a TR approach using the Maia platform) and Treatment as Usual (15 sessions of multimedia content of educational/rehabilitation activities delivered via telemedicine platfom). It expected that the TR system to be considered acceptable in terms of efficiency (usability and acceptability of the technologies) and clinically effective, with positive impacts on both quality of life and central and peripheral functioning in these patients.

ELIGIBILITY:
Inclusion Criteria:

* Adult subjects (>18 years old) with central and/or peripheral neurotoxic sequelae following a history of cancer treated with chemotherapeutic agents (Cisplatin and Taxanes), in accordance with the criteria of the International Cognitive Cancer Task Force (Wefel et al., 2011. 10.1016/S1470-2045(10)70294-1)
* agreement to participate with the signature of the informed consent form;

Exclusion Criteria:

* Ongoing chemotherapy treatment;
* Pre-existing neurological or psychiatric comorbidities (e.g., epilepsy, post-stroke disability, neurodegenerative diseases, genetically based polyneuropathy);
* Severe visual or hearing impairments that could interfere with the use of technology;
* Severe cognitive impairment (Mini-Mental State Examination score <18);
* Severe postural disability associated with a high risk of falling at home, as documented in the clinical evaluation;
* Contraindications to undergoing MRI examination;
* Ongoing rehabilitation treatment.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2025-09-01 (Estimated); Primary Completion 2026-07-31 (Estimated); Study Completion 2026-08-31 (Estimated)

PRIMARY OUTCOMES:
Changes in Activation level of Patients measured by Patient Activation Measure 13 (PAM13; Hibbard et al., 2004) | Time Frame: Baseline, post-treatment (up to 5 weeks)
  PAM13 is a 13-item scale that assesses a person's underlying knowledge, skills and confidence integral to managing his or her health and healthcare. PAM13 total score ranging from 0 to 100. Higher values represent a better outcome. Specifically, individuals in the lowest activation level do not yet understand the importance of their role in managing their health and have significant knowledge gaps and limited self-management skills. Individuals in the highest activation level are proactive with their health, have developed strong self- management skills, and are resilient in times of stress or change.

SECONDARY OUTCOMES:
Change in Functional Assessment of Cancer Therapy-Cognitive Function - FACT-Cog (Fardell et al., 2022. 10.1002/pon.5928); | Baseline, post-treatment (up to 5 weeks)
  FACT-Cog is a 37 item self-report tool on 5-point Likert scale to assess perceived cognitive function in adult cancer patients with chemotherapy-induced cognitive problems
Change in EORTC CIPN-20 questionnaire (Postam et al., 2005). | Baseline, post-treatment (up to 5 weeks)
  EORTC CIPN-20 is a 20-item self-report questionnaire to assess patients' experience of symptoms and functional limitations related to chemotherapy-induced peripheral neuropathy;
Change in Patient Health Engagement Scale (PHE) (Graffigna et al., 2017) | Baseline, post-treatment (up to 5 weeks)
  Patient Health Engagement Scale (PHE-s) is a validated tool designed to measure a person's level of engagement in managing their own health, based on the Patient Health Engagement (PHE) Model.
Change in global cognitive functioning and subdomains measured by Montreal Cognitive Assessment (MoCA; Santangelo et al., 2015) | Baseline, post-treatment (up to 5 weeks)
  MoCA is a screening test for global cognitive functioning. It includes tasks involving several domains: visuospatial/executive function tests, naming, selective and sustained attention, language, abstraction, memory and orientation. High scores are indicative of better general cognitive performance.
Change in visuoperceptual and attentional abilities measured by Trail Making Test (TMT part-A and part-B; Giovagnoli et al., 1996) | Baseline, post-treatment (up to 5 weeks)
  TMT is a neuropsychological test that involves visual scanning (TMT-A) and dual-task (TMT-B). The TMT is scored by how long it takes to complete each part of the test. High execution times indicate poor performance.
Change in long term visual memory measured by Free and Cued Selective Reminding Test (FCSRT) (Frasson et al., 2011) | Baseline, post-treatment (up to 5 weeks)
  FCSRT is a visual memory test that maximises encoding specificity. It assesses learning (immediate recall) and visual long-term (delayed recall) memory of visual stimuli. The administration is divided into three phases: 1) Encoding phase: naming of stimuli (three boards with four coloured stimuli each) and verification of encoding with cue; 2) Immediate recall phase: free immediate recall + recall with a cue for not recalled stimuli (this sequence is repeated three times with interference task between trials); 3) deferred recall phase (after 30 minutes of non-verbal tasks): free deferred recall + recall with a cue for not recalled stimuli. Six scores can be obtained: Immediate Free Recall (spontaneous recall in the three trials; range 0-36); Immediate Total Recall (total recall in the three trials - range 0-36); Delayed-Free Recall (range 0-12); Delayed Total Recall (range 0-12); Index of Sensitivity of Cueing (ISC) and Number of intrusions. Higher scores indicate better performance.
Change in Static and dynamic balance measured by Mini-Best Test (Franchignoni et al., 2010) | Baseline, post-treatment (up to 5 weeks)
  The Mini-BESTest aims to identify the disordered systems underlying the postural control responsible for poor functional balance. This tool is composed by 27 tasks (36 items in total) assessing bio-mechanical constraints, stability limits/verticality, anticipatory responses, postural responses, sensory orientation, and stability in gait. Each item is scored based on ordinal scale scoring from 0- 3 where 3 = best performances and 0 = worst performances. The total score is provided as a percentage. Higher scores are indicative of better performance.
Change in Aerobic Capacity and Gait measured by 6' Minute Walking Test (6MWT) | Baseline, post-treatment (up to 5 weeks)
  6' Minute Walking Test (6MWT) has been validated as a general indicator of overall physical performance and mobility for older people (Duncan et al 1993; Harad et al 1999). The total distance walked is measured.
Change in strength level using a dynamometer | Baseline, post-treatment (up to 5 weeks)
  dynamometer

OTHER OUTCOMES:
Changes in brain morphometry as detected by Magnetic Resonance Imaging Examination. | Baseline, post-treatment (up to 5 weeks)
  T1-3D MPRAGE, FLAIR 3D and T2 will be collected to test changes in brain morphometry
Changes in structural connectivity as detected by Magnetic Resonance Imaging Examination. | Baseline, post-treatment (up to 5 weeks)
  DWI sequences will be collected to detect changes in structural connectivity
Changes in functional connectivity as detected by Magnetic Resonance Imaging Examination. | Baseline, post-treatment (up to 5 weeks)
  Resting-State fMRI (Multi echo - Multi-Band) and EPI-T2* images will be collected for the assessment of brain activity at rest and functional connectivity.
Changes in muscle tissue inflammation as detected by Magnetic Resonance Imaging Examination. | Baseline, post-treatment (up to 5 weeks)
  T2 mapping (T2 SE multi-echo) will be collected to measure change in inflammation
Changes in muscle fiber integrity as detected by Magnetic Resonance Imaging Examination. | Baseline, post-treatment (up to 5 weeks)
  Muscle diffusion tensor imaging (DWI-STE) will be collected to measure muscle fiber integrity
Changes in fat fraction as detected by Magnetic Resonance Imaging Examination. | Baseline, post-treatment (up to 5 weeks)
  Multi-point Dixon (6-point multi-echo GRE Dixon) will be collected to evaluate fat fraction.
Changes in inflammatory and anti-inflammatory cytokines as measured by blood sampling | Baseline, post-treatment (up to 5 weeks)]
  The sera will be collected, centrifuged, stored, frozen at -80 C degrees, and shipped (when necessary) to the chosen sample-processing center. The serum will be used to measure by Enzyme-Linked ImmunoSorbent Assay (ELISA) and by Automated Immunoassay System (ELLA) the Inflammatory cytokines (TNF, IL1beta, TGF-beta, IL-6), and Anti-inflammatory cytokines (IL-10).
Changes in neurotrophic and neuroendocrine factors as measured by blood sampling | Baseline, post-treatment (up to 5 weeks)]
  The sera will be collected, centrifuged, stored, frozen at -80 C degrees, and shipped (when necessary) to the chosen sample-processing center. The serum will be used to measure by Enzyme-Linked ImmunoSorbent Assay (ELISA) and by Automated Immunoassay System (ELLA) the neurotrophic and neuroendocrine factors such as Brain-derived neurotrophic factor (BDNF), neurofilaments and neurotransmitters (acetylcholine, noradrenaline, and adrenaline), cortisol, VEGF, IGF-1 and irisin.

CONTACTS AND LOCATIONS:
Overall Officials: Francesca Baglio, Principal Investigator — IRCCS Fondazione Don Carlo Gnocchi ONLUS
Locations (1):
- IRCCS Fondazione Don Carlo Gnocchi ONLUS, Milan, Italy

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: internet page of Institution — http://www.dongnocchi.it/ricerca-scientifica/i-centri-irccs/irccs-s-maria-nascente-milano/caditer
- See also: internet page of Research Unit — http://caditer.dongnocchi.it/